CLINICAL TRIAL: NCT01151397
Title: Does 3 Months Therapy With Vitamin D + Peg + Ribavirin Improve SVR in Genotype 2,3 Chronic Hepatitis C Patients?
Brief Title: Does 3 Months Therapy With Vitamin D + Peg + Ribavirin Improve Sustained Virologic Response (SVR) in Genotype 2, 3 Chronic Hepatitis C Patients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Liver Clinic, Ziv medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Genotype 2,3 HCV +Vitamin D
Record Dates: First submitted 2010-06-16; First posted 2010-06-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Hepatitis C
Keywords: SVR; VITAMIN D; Hepatitis C; Genotype 2,3; Naive; RVR
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Polyethylene Glycols; Vitamin D; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peg + Vitamin D + Ribavirin (Active Comparator): Peg + Vitamin D + Ribavirin for 3 months
  Interventions: Drug: Peg + Vitamin D + Ribavirin
- Peg + Ribavirin (Active Comparator): Peg + Ribavirin for 6 months
  Interventions: Drug: Peg + Ribavirin

INTERVENTIONS:
Drug: Peg + Vitamin D + Ribavirin — Peg+ Vitamin D+ Ribavirin for 3 months
  Arms: Peg + Vitamin D + Ribavirin
Drug: Peg + Ribavirin — Peg+ Ribavirin for 6 months
  Arms: Peg + Ribavirin

SUMMARY:
Standard therapy for chronic hepatitis C virus (HCV) is (Peg/RBV) combination therapy obtaining sustained virologic response (SVR) in 80% of naïve patients with genotype 2,3. Studies rarely address the issues of improving host factors. The current study examines

1. Does 3 months therapy with Vitamin D+ Peg + Ribavirin could improve viral response and shorten treatment duration (from 24 weeks to 12 weeks)
2. whether Vitamin D levels predicts negative treatment outcome.

DETAILED DESCRIPTION:
Standard therapy for chronic hepatitis C virus (HCV) is (Peg/RBV) combination therapy obtaining sustained virologic response (SVR) in 80% of naïve patients with genotype 2, 3. Studies rarely address the issues of improving host factors. The current study examines whether adding vitamin D, a potent immunomodulator, for 3 months therapy could improve viral response. The working hypothesis is that 3 months therapy with Vitamin D + Peg + Ribavirin significantly improves RVR, EVR, and SVR.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* chronic genotype 2,3 HCV infection
* treatment Naive negative sero for HBV, HDV and HIV viral infections
* absolute neutrophil count of >1500 per cubic millimeter
* a platelet count of >90,000 per cubic millimeter normal hemoglobin level

Exclusion Criteria:

* decompensated liver disease (cirrhosis with CP score >9)
* another cause of clinically significant liver disease hepato cellular carcinoma
* psychiatric Disorder
* chronic heart failure
* pregnant women
* uncontrolled diabetes with retinopathy Arrhythmia Active CAD
* positive sero for HBV, HDV and HIV viral infections or other autoimmune liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-02 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
sustained virologic response (SVR)rate | 24 weeks
  the SVR rate data will be collected and compared for 2 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv medical center liver unit, Safed, Israel, Israel